CLINICAL TRIAL: NCT07252830
Title: Identification of Asymptomatic Patients at Very High Cardiovascular Risk: Contribution of a Strategy Based on Carotid and Coronary Explorations, Compared to Simple Risk Calculation Using the European "SCORE 2" Algorithm.
Brief Title: Identification of Asymptomatic Patients at Very High Cardiovascular Risk: Contribution of a Strategy Based on Carotid and Coronary Explorations, Compared to Simple Risk Calculation Using the European "SCORE 2" Algorithm. (IDEA-CVR)
Acronym: IDEA-CVR
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Collaborators: Polyclinique Poitiers (Unknown)
Responsible Party: Sponsor
Other Study IDs: IDEA-CVR
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; Atheroma; Cholesterol; Cardiovascular (CV) Risk
MeSH Terms: conditions — Myocardial Infarction; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic patients, in screening / primary prevention
  Interventions: Other: SCORE2

INTERVENTIONS:
Other: SCORE2 — the European algorithm "SCORE 2", available online (figure 1). It allows the calculation of the absolute risk in % of occurrence of a fatal or non-fatal CV event (myocardial infarction, stroke) over 10 years.

SUMMARY:
To prevent myocardial infarction ( MI), coronary atheroma development by LDL-cholesterol deposition in the arterial wall is the basis. Since atheromatous plaques develop slowly before becoming symptomatic, their early detection in asymptomatic patients and the implementation of an effective strategy to prevent their progression constitute the most promising primary prevention strategy. In younger subjects, the main modifiable pro-atheromatous factors are smoking and an excessively high LDL-C level, partly genetically predetermined, but also favored by a diet too rich in saturated fats and a lack of physical activity. In the French national MI registry, the average age of patients is 62 years (Arch Cardiovasc Dis 2021 Oct;114(10):647-655). Half of MIs therefore occur at working age due to rupture of atheromatous plaques, which had developed during the months/years preceding the acute event.

According to the latest recommendations of the European Society of Cardiology (ESC) on CV prevention published in August 2021, the visualization of coronary or carotid atheromatous plaques justifies considering the patient as having atherosclerotic cardiovascular disease (ASCVD), and automatically places them in the "very high CV risk" category, with an LDL-cholesterol target of <0.55 g/L. However, these recommendations do not clearly define the criteria justifying the use of imaging in asymptomatic patients.

In current practice, CV risk stratification for asymptomatic patients with no prior CV disease is currently based on risk calculation using the European "SCORE 2" algorithm, available online. It allows the calculation of the absolute risk in % of occurrence of a fatal or non-fatal CV event (myocardial infarction, stroke) over 10 years.

The main objective of this study is to describe patients reclassified as "very high CV risk" following the detection of atheroma plaques formed in relation to their risk level estimated by SCORE2.

DETAILED DESCRIPTION:
It is a national, single-center, retrospective and prospective study on the collection of routine care data.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years and < 80 years referred to general cardiology consultation
* LDL-C level > 1.6 g/L, or LDL-C level > 1.3 g/L with at least one associated major cardiovascular (CV) risk factor (RCF) (smoking, hypertension, diabetes).
* Coronary artery reserve assessment and EDTSA performed in a day hospital

Exclusion Criteria:

* Known or suspected carotid atherosclerotic disease
* Significant ischemic heart disease known or suspected at the time of the initial consultation
* Protected adult patient (patient under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative decision)
* Opposition expressed by the patient to the use of their health data.
* Patient may have limited understanding of the information sheet

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology team of the Poitiers polyclinic (France)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Very high risk cardiovascular (yes/no) | 12 months
  Patients reclassified as "very high CV risk" (Yes/No) compared to the risk level estimated by SCORE2.
  SCORE2 is determined by an online calculator from the European Society of Cardiology (ESC).

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinqiue de Poitiers, Poitiers, France